CLINICAL TRIAL: NCT00300976
Title: (Intervention Study) A Randomized Controlled Study of the Intensive Therapy and the Conventional Therapy for the Suppression of the Vascular Complications in the Type 2 Diabetic Patients (Follow-up Study) A Randomized Controlled Study Comparing Intensive Therapy and Conventional Therapy in the Reduction of Vascular Complications in Type 2 Diabetic Patients: A Follow-up Study After Intervention
Brief Title: The Japan Diabetes Optimal Integrated Treatment Study for 3 Major Risk Factors of Cardiovascular Diseases
Acronym: J-DOIT3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Japan Foundation for the Promotion of International Medical Research Cooperation (Other)
Collaborators: Japan Diabetes Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J-DOIT3
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2
Keywords: Blood glucose; Blood pressure; Lipids
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: (Intervention study) A multi-center, open-label, randomized controlled study, which compared the efficacy of intensive therapy and conventional therapy in type 2 diabetic patients
  (Follow-up study) A prospective cohort study with a 5-year long-term follow-up period
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive therapy (Experimental)
  Interventions: Behavioral: Lifestyle consultation: weight control, diet, exercise
- Conventional therapy (Active Comparator)
  Interventions: Behavioral: Lifestyle consultation: weight control, diet, exercise

INTERVENTIONS:
Behavioral: Lifestyle consultation: weight control, diet, exercise — Behavioral: Lifestyle modification including weight control, with the goal of BMI 22.
  Drug: Drugs are added in a stepwise manner to control blood glucose, blood pressure and lipid metabolism, using mainly hypoglycemic drugs, ACEI/ARB and statins, respectively. Management goals are: HbA1c < 6.2%, BP < 120/75 mmHg, HDL-C 40 mg/dL , LDL-C < 80 mg/dL, TG < 120 mg/dL.
  Follow-up study (Not provided)
  Arms: Intensive therapy
Behavioral: Lifestyle consultation: weight control, diet, exercise — Behavioral and Drug: The physician in charge is to administer appropriate therapy in accordance with the Guidelines.
  Follow-up study (Not provided)
  Arms: Conventional therapy

SUMMARY:
(Intervention study) The objective of the study is to confirm the superiority of the intensive therapy to the conventional therapy concerning the prevention of the incidence or exacerbation of vascular complications caused by diabetes mellitus (DM) by a randomized controlled study in patients with type 2 DM.

(Follow-up study) The objective of the follow-up study is to evaluate the long-term efficacy of intensive versus conventional therapy in the effect on mortality and the prevention of the incidence or exacerbation of vascular complications caused by diabetes mellitus through a post-intervention follow-up research conducted after the multi-center, open-label, randomized parallel-group study comparing the efficacy of intensive versus conventional therapy in type 2 diabetic patients.

DETAILED DESCRIPTION:
(Intervention study) The objective of the study is to confirm the superiority of the intensive therapy to the conventional therapy concerning the prevention of the incidence or exacerbation of vascular complications caused by diabetes mellitus by a randomized controlled study in patients with type 2 DM. The primary outcome measure is occurrence of myocardial infarction, coronary bypass surgery, percutaneous transluminal coronary angioplasty, stroke, carotid endarterectomy, percutaneous transluminal cerebral angioplasty, carotid artery stenting, or death.

(Follow-up study) The objective of the follow-up study is to evaluate the long-term efficacy of intensive versus conventional therapy in the effect on mortality and the prevention of the incidence or exacerbation of vascular complications caused by diabetes mellitus through a post-intervention follow-up research conducted after the multi-center, open-label, randomized parallel-group study comparing the efficacy of intensive versus conventional therapy in type 2 diabetic patients. The primary endpoint is identical to that in the intervention study. In addition, overall survivalall-cause mortality will be evaluated as a key secondary endpoint.

ELIGIBILITY:
(Intervention study)

Inclusion Criteria:

Subjects were considered eligible if they were 45 years old or older but younger than 70 years old at study entry, had type 2 diabetes and met both "(1) and (2)" or both "(1) and (3)" described below. [Note: Those who met all three "(1), (2) and (3)" were also considered eligible for inclusion.](1) Glycemic control Those with HbA1c 6.9% or greater despite treatment with any of the three regimens given below. Diet and exercise therapy alone, Diet and exercise therapy plus 1 oral anti-diabetic drug, Diet and exercise therapy plus, GI and 1 other oral anti-anti-diabetic drug (2) Blood pressure control Those with the following casual blood pressure (BP) level as measured on an outpatient basis, Systolic BP 140 mmHg or diastolic BP 90 mmHg while not on an antihypertensive agent, Systolic BP 130 mmHg or diastolic BP 80 mmHg while on 1 or 2 ARB, ACEI or long-acting CCB Those receiving antihypertensive agents other than ARB, ACEI or long-acting CCB were not eligible for study entry, with the exception of those who were receiving these agents for other purposes than blood pressure lowering. (3) Lipid metabolism Those with the following fasting lipid levels while not on a lipid-lowering agent LDL-cholesterol, 120 mg/dL (as calculated by using the Friedewald formula) Triglycerides, 150 mg/dL HDL-cholesterol, < 40 mg/dL Subjects receiving 1 lipid-lowering agent were judged eligible for study entry if they met any of the above criteria. However, care needs to be taken to ensure that those on fibrates discontinue the fibrate treatment at the start of the study when they are assigned to the intensive therapy arm.

Exclusion Criteria:

1. Those with poorly controlled hypertension despite pharmacological therapy (systolic BP 200 mmHg or diastolic BP 120 mmHg) 2. Those on insulin therapy 3. Those with non-diabetic renal disease 4. Those in whom type 1 and other diabetes due to pathogenic mechanisms other than those associated with type 2 diabetes is strongly suspected 5. Those who tested anti-GAD antibody*-positive 6. Those with LDL-cholesterol 200 mg/dL 7. Those suspected of having secondary hypertension other than renal parenchymal hypertension 8. Those suspected of having hereditary lipid disorder with a strong family history of lipid metabolic disorder 9. Those who were receiving antihypertensive agents other than ARB, ACEI, long-acting CCB, except where they were receiving these agents for other purposes than blood pressure lowering 10. Those who were receiving 3 or more antihypertensive agents (i.e., ARB, ACEI, and long-acting CCB), except where they were receiving these agents for other purposes than blood pressure lowering 11. Those with more serious retinopathy than proliferative retinopathy 12. Renal failure (serum Cr: 2.0 mg/dL in men; 1.5 mg/dL in women) 13. Those with a history of cardiac failure or those with cardiac failure 14. Those who were pregnant or potentially pregnant 15. Those who met any of the following criteria and who had BNP 100 pg/mL, Myocardial infarction, Angina pectoris (or a history of disease), History of coronary artery bypass graft (CABG), History of percutaneous coronary angioplasty (PTCA), Other cardiac disease, ECG findings of left ventricular hyperplasia, Abnormal ECG findings (excluding isolated extrasystole or right bundle branch block [RBBB]) 16. Those judged by the physician in charge to be ineligible for study entry

(Follow-up study)

Inclusion criteria:

Of the subjects in the randomized controlled study comparing intensive therapy and conventional therapy in type 2 diabetic patients (J-DOIT3), those who provide written informed consent to participate in the follow-up study will be enrolled regardless of completion or discontinuation from the randomized controlled study (If the subject is unable to provide informed consent for any reason, consent from his/her legal representative is allowed).

Exclusion criteria:

A subject who is assessed as ineligible by the investigator will be excluded from the follow-up study

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2542 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The occurrence of myocardial infarction, coronary bypass surgery, percutaneous transluminal coronary angioplasty, stroke, carotid endarterectomy, percutaneous transluminal cerebral angioplasty, carotid artery stenting, or death | Every 12 months, at the end of the study.

SECONDARY OUTCOMES:
Occurrence of myocardial infarction, stroke or death | Every 12 months, at the end of the study.
Onset or progression of nephropathy | Every 6 months, at the end of the study.
Lower limb vascular events (amputation or revascularization of lower limb) | Every 12 months, at the end of the study.
Onset or progression of retinopathy | Every 12 months, at the end of the study.
All-cause mortality (deaths due to any cause) | Every 12 months, at the end of the study.
  This measure is only evaluated with follow-up study.

OTHER OUTCOMES:
Development of severe hypoglycemia (requiring assistance from another person and/or hospitalization) | Every 12 months, at the end of the study.
  This measure is only evaluated with follow-up study.
Hospitalization for heart failure | Every 12 months, at the end of the study.
  This measure is only evaluated with follow-up study.
Development of malignant neoplasms | Every 12 months, at the end of the study.
  This measure is only evaluated with follow-up study.
Occurrence of fractures | Every 12 months, at the end of the study.
  This measure is only evaluated with follow-up study.
Changes in cognitive function (MMSE) | At the end of the study.
  This measure is only evaluated with follow-up study.
Changes in QOL (EQ-5D) | At the enrollment, at the end of the study.
  This measure is only evaluated with follow-up study.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Principal Investigator — Tokyo University
Locations (1):
- The University of Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Sasako T, Ueki K, Miyoshi K, Miyake K, Aoyama T, Okazaki Y, Ishizuka N, Yamauchi T, Noda M, Kadowaki T; J-DOIT3 Study Group. Effect of a Multifactorial Intervention on Retinopathy in People With Type 2 Diabetes: A Secondary Analysis of the J-DOIT3 Randomized Clinical Trial. JAMA Ophthalmol. 2025 Dec 1;143(12):989-997. doi: 10.1001/jamaophthalmol.2025.3819. PMID 41129145
- [Derived] Sasako T, Ueki K, Miyake K, Okazaki Y, Takeuchi Y, Ohashi Y, Noda M, Kadowaki T. Effect of a Multifactorial Intervention on Fracture in Patients With Type 2 Diabetes: Subanalysis of the J-DOIT3 Study. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2116-e2128. doi: 10.1210/clinem/dgab013. PMID 33491087
- [Derived] Ueki K, Sasako T, Okazaki Y, Kato M, Okahata S, Katsuyama H, Haraguchi M, Morita A, Ohashi K, Hara K, Morise A, Izumi K, Ishizuka N, Ohashi Y, Noda M, Kadowaki T; J-DOIT3 Study Group. Effect of an intensified multifactorial intervention on cardiovascular outcomes and mortality in type 2 diabetes (J-DOIT3): an open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2017 Dec;5(12):951-964. doi: 10.1016/S2213-8587(17)30327-3. Epub 2017 Oct 24. PMID 29079252
- [Derived] Ueki K, Sasako T, Kato M, Okazaki Y, Okahata S, Katsuyama H, Haraguchi M, Morita A, Ohashi K, Hara K, Morise A, Izumi K, Ohashi Y, Noda M, Kadowaki T; J-DOIT3 Study Group. Design of and rationale for the Japan Diabetes Optimal Integrated Treatment study for 3 major risk factors of cardiovascular diseases (J-DOIT3): a multicenter, open-label, randomized, parallel-group trial. BMJ Open Diabetes Res Care. 2016 Jan 25;4(1):e000123. doi: 10.1136/bmjdrc-2015-000123. eCollection 2016. PMID 26843962